CLINICAL TRIAL: NCT07225959
Title: A Phase 2, Open-Label, Long-Term Study to Evaluate the Safety, Pharmacokinetics, and Occurrence of Anti-Drug Antibodies in Healthy Participants Following Annual Doses of CD388, a Novel Long-Acting Antiviral Conjugate
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Occurrence of Anti-Drug Antibodies Following Annual Doses of CD388
Acronym: NAVIGATE-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cidara Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CD388.SQ.2.07
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: Influenza; Antiviral Agents
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD388 (Experimental): Each participant will receive a single 450 mg dose of CD388 by subcutaneous (SQ) injection followed 1 year later by a repeat single 450 mg dose of CD388 administered by SQ injection.
  Interventions: Combination Product: CD388 Injection

INTERVENTIONS:
Combination Product: CD388 Injection — CD388 liquid for injection

SUMMARY:
The goal of this clinical study is to learn if giving repeated annual doses of the experimental drug CD388 is safe and how the body reacts to it in healthy adults who have already received one dose without serious side effects. The study aims to determine if the body makes antibodies against CD388 after repeated doses, which might affect how the drug works or how safe it is, and to better understand the safety and tolerability of repeated doses. Participants will receive two doses of CD388 over two years and be monitored for 18 months. Researchers will check for immune responses against the drug, watch for any side effects, and measure how the drug behaves in the body over time. This study is based on the idea that people who tolerated CD388 well before will likely continue to tolerate it safely with repeated annual dosing, and that the risk of immune reactions will remain low. Expanded access to the study drug will not be provided to participants after the study ends.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, long-term study to evaluate the occurrence of anti-drug antibodies (ADAs) directed to CD388 during an 18-month period following administration of 2 annual doses of CD388 in healthy participants who previously completed study CD388.SQ.2.05, having received a dose of the active drug without experiencing any serious adverse event(s) (SAE[s]) during that study. This study will also evaluate the safety and tolerability of CD388 and the pharmacokinetics (PK) of CD388 following repeated annual dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent and comply with scheduled visits, laboratory tests, and other study procedures.
2. Be a male or female adult aged 18 to 66 years of age who previously completed participation in Study CD388.SQ.2.05, having received a SQ CD388 dose of either 150 mg, 300 mg or 450 mg. (Note: Participants in this study may have received seasonal influenza vaccine prior to enrollment in this study and may receive influenza vaccine during this study, with certain exceptions as described in the protocol.)
3. Be in stable health at the time of screening and enrollment (in the Investigator's clinical judgment). Participants may not have a history of underlying hematologic, oncologic, renal, autoimmune, cardiac, or pulmonary conditions; or be considered at risk of developing complications from influenza infection per the United States Centers for Disease Control and Prevention (CDC) guidelines (chronic obstructive pulmonary disease [COPD], asthma, current immune-compromised cancer [except non-melanomatous skin cancer], or diabetes). Study participants will be included based on medical history and vital signs obtained during the screening process.
4. Have a body mass index (BMI; calculated as weight in kilograms [kg] divided by height in meters [m] squared)) of ≥18 kg/m^2.
5. Must agree to the following contraception requirements:

   a. Females of childbearing potential must use a highly effective, preferably user-independent, method of contraception (failure rate of less than 1 percent per year when used consistently and correctly) from ≥2 weeks prior to enrollment and agree to remain on a highly effective method from Day 1 until 40 weeks after each study intervention administration, the end of relevant systemic exposure. Note: A female is considered of childbearing potential (i.e., fertile) following menarche and until becoming postmenopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in females not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

   Note: Contraceptive (birth control) use by participants should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies.
6. Must agree not to donate blood from Day 1 until 40 weeks after each administration of CD388.
7. Must be able to read, understand, and complete protocol questionnaires using the Sponsor-designated diary mode (eDiary or paper) and language, and be willing and able to adhere to the prohibitions and restrictions specified in this protocol. If eDiary is designated, the participant must be able to use a smartphone/tablet/computer. If an appropriate language version is not available in either eDiary or paper, the participant must not be enrolled. The diary mode and approved languages will be designated by the Sponsor prior to study start.
8. Must be willing to provide verifiable identification, has means to be contacted, and is able to contact the Investigator/study site and communicate reliably during participation in this study.

Exclusion Criteria:

1. Have a known or suspected allergy or history of anaphylaxis or other serious adverse reactions to zanamivir (following administration of inhaled or intravenous formulations), monoclonal antibodies (including crystallizable fragment [Fc] domains), or any of the components of CD388.
2. Have an acute illness (including acute respiratory illnesses) or body temperature ≥38.0 degrees Celsius (ºC) (≥100.4 degrees Fahrenheit [ºF]) within 7 days prior to each administration of CD388. (Note: Enrollment and/or receipt of study intervention at a later date, subsequent to resolution of the illness [within the screening period], is permitted.)
3. Have a serious and/or clinically unstable condition, including but not limited to, a psychiatric condition including recent (within the past year) or active suicidal ideation/behavior, Alzheimer's disease, or any other condition which in the opinion of the Investigator might lead to hospitalization or death within this study period and for which enrollment would not be in the participant's best interest, or could prevent, confound, or limit the protocol-specified assessments.
4. Have any history of alcohol or substance abuse which in the opinion of the Investigator might interfere with conduct of this study as planned.
5. Had major surgery (e.g., cardiac, pulmonary, neurologic, or abdominal operations) within 4 weeks prior to screening, or will not have fully recovered from such prior surgery; or has major surgery planned during the time the participant is expected to participate in this study.
6. Had screening electrocardiogram (ECG) findings of prolonged QT interval corrected using Fridericia's formula (QTcF) (greater than 450 milliseconds [msec] in males or greater than 470 msec in females), prolonged PR interval (greater than 220 msec), second- or third-degree heart block, or other clinically significant dysrhythmia.
7. Have any finding (at the time of screening) that may significantly increase the risk of participation in this study, affect the ability to participate in this study, or impair interpretation of the study data.
8. Have current or planned participation in another clinical study where study intervention is being administered while participating in this current study. Note: Concurrent enrollment is allowed during the follow-up phase of the other clinical study or in case the study intervention in the other clinical study is a marketed product already approved for another indication - exception being if the other study requires study interventions that could affect the safety assessments of this present study (e.g., clinical laboratory tests).
9. Have received any experimental drug, vaccine, or biologic agent within the past 90 days or 5 half-lives (whichever is longer) prior to study intervention administration.
10. Have a contraindication to SQ injections and venipunctures (e.g., bleeding disorders).
11. Have donated ≥450 mL of blood product (1 unit) for any reason within 30 days of screening or have plans to donate blood product during the study.
12. Are currently pregnant or breastfeeding, intends to become pregnant or breastfeed, or has a positive pregnancy test during the screening period.
13. Has direct involvement in the proposed study or other studies under the direction of the Investigator, sub-investigators, or study site personnel; is a family member of an individual with such direct involvement; or is an employee of the Sponsor.
14. Did not complete participation in protocol CD388.SQ.2.05, or experienced an SAE during that study, or was enrolled in CD388.SQ.2.05 despite not meeting that study's eligibility (one or more Inclusion Criteria not met or one or more Exclusion Criteria met), as determined on retrospective review, irrespective of completion status.
15. In the opinion of the Investigator, is unlikely to adhere to the requirements of this study.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Anti-Drug Antibodies (ADAs) in Participants Administered CD388 | On Day 1 (pre-dose baseline), Day 29, Day 85, Day 169, and Day 197 in Study Period 1; on Day 1 (pre-dose), Day 29, Day 85, Day 169, and Day 197/End of Study (EOS) in Study Period 2
  Evaluation of blood serum samples for the occurrence of treatment-emergent anti-drug antibodies (ADAs) or treatment-boosted ADAs (based on an increase in ADA titer in samples positive for ADA at baseline) directed to CD388 in participants following administration of each annual dose of CD388.

SECONDARY OUTCOMES:
Incidence and Severity of Treatment-Emergent Adverse Events (TEAEs) after Administration of Study Drug | From Study Period 1 Day 1 after study drug dosing through Study Period 2 Day 197/EOS
  Safety and tolerability of CD388 will be evaluated by assessing the number of participants with incidences of TEAEs following the administration of study drug. TEAEs include but are not limited to adverse events (AEs), serious adverse events (SAEs), injection site reactions (ISRs), and any potentially clinically significant changes from baseline seen in vital signs and clinical laboratory parameters.
Plasma Concentrations at Specified Timepoints Following Administration of CD388 | In both Study Periods 1 and 2 on Day 1 (pre-dose), Day 8, Day 29, Day 85, Day 169, and Day 197/EOS as applicable
  Evaluation of the plasma concentration of CD388 at specified timepoints after study drug dosing.
Trough Plasma Concentration at 24 Weeks (C[trough24w]) Following Administration of CD388 | In both Study Periods 1 and 2 on Day 169
  Evaluation of the trough plasma concentration at 24 weeks (C[trough24w]) after study drug dosing.
Maximum Plasma Concentration (C[max]) Following Administration of CD388 | In both Study Periods 1 and 2 on Day 1 (pre-dose), Day 8, Day 29, Day 85, Day 169, and Day 197/EOS as applicable
  Evaluation of the maximum plasma concentration (C[max]) after study drug dosing.
Area Under the Plasma Concentration-Time Curve (AUC) Following Administration of CD388 | In both Study Periods 1 and 2 on Day 1 (pre-dose), Day 8, Day 29, Day 85, Day 169, and Day 197/EOS as applicable
  Evaluation of the area under the plasma concentration-time curve (AUC) after study drug dosing.
Correlation of Plasma Concentration of CD388 and Titer of Anti-CD388 Antibodies at Time Points Where ADAs are Present | In both Study Periods 1 and 2 on Day 1 (pre-dose), Day 29, Day 85, Day 169, and Day 197/EOS as applicable
  Comparison of the plasma concentration of CD388 to the titer of CD388 ADAs at time points where ADAs are present in participants administered CD388.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Davarpanah, MD, JD, Study Director — Cidara Therapeutics Inc.
Locations (3):
- United States (2):
  - Floridian Clinical Research, Miami Lakes, Florida
  - Spartanburg Medical Research, Spartanburg, South Carolina
- hVIVO Serviced Limited, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No